CLINICAL TRIAL: NCT04299204
Title: Which Factor Affect the Success of Pediatric PCNL?: Single Center Experiences, Over 20 Years: Cohort Study
Brief Title: The Success of Pediatric Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Government Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: OsmaniyeGH
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Nephrolithiasis
Keywords: Urolithiasis; Pediatrics; Percutaneous
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Intervention Model Description: the data into two groups. In group-1, PCNL was performed in the first 10 years period (1997-2007); in group-2, PCNL was performed in the second ten years period from 2008 to the present.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Years 1997-2007 (Experimental): Group-1, PCNL was performed in the first 10 years period (Years 1997-2007);
  Interventions: Procedure: Percutaneous nephrolitotomy
- 2008- to the present (Experimental): The PCNL was performed in the second ten years period from 2008 to the present.
  Interventions: Procedure: Percutaneous nephrolitotomy

INTERVENTIONS:
Procedure: Percutaneous nephrolitotomy — Pediatric PCNL

SUMMARY:
Between June 1997-June 2018, 573 pediatric patients underwent PCNL for renal stone disease by senior surgeons. Data was disunited into 2 groups.

The study showed that PCNL is an operator-dependent procedure, with the improvement of outcomes over time, presumably due to increased operator experience and the involvement of a team member with substantial prior experience During 20 years, by gaining experience and with the development of new tools and optics, fluoroscopy time, operation time, blood loss and complication rates decreased and stone-free rates increased.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with kidney stone

Exclusion Criteria:

* Patients with a solitary kidney

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 553 (Actual)
Dates: Start 1998-01-15 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of clinical experience of Percutaneous nephrolitotomy | over 20 years
  The duration of clinical experience affects complication rates, success rates. Intraoperative and postoperative data was contained, preoperative and postoperative GFR (calculated with Cockcroft Gault equations), changing hemoglobin levels, transfusion rate, complications according to the Clavien classification.

SECONDARY OUTCOMES:
Changing of complications managements | Over 20 years
  Rate of and changing of Management of complications in pediatric patients

IPD SHARING:
Plan to Share IPD: Undecided
The data belonged to Cukurova University, Department of Urology

REFERENCES:
- [Result] Citamak B, Altan M, Bozaci AC, Koni A, Dogan HS, Bilen CY, Sahin A, Tekgul S. Percutaneous Nephrolithotomy in Children: 17 Years of Experience. J Urol. 2016 Apr;195(4 Pt 1):1082-7. doi: 10.1016/j.juro.2015.11.070. Epub 2015 Dec 9. PMID 26682755